CLINICAL TRIAL: NCT00410605
Title: Phase II Trial of Bevacizumab Combined With Lenalidomide and Dexamethasone (BEV/REV/DEX) in Relapsed or Refractory Multiple Myeloma
Brief Title: Bevacizumab, Lenalidomide, and Dexamethasone in Patients With Relapsed or Refractory Stage II or III Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00150; NCI-2009-00150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); H-2006-0269 (Other: UW Health Sciences IRB); CDR0000521546; HO06401 (Other: University of Wisconsin Hospital and Clinics); 7313 (Other: CTEP); U01CA062491 (NIH); P30CA014520 (NIH); NCT00406328 (obsolete NCT alias)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma in Relapse; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bevacizumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, oral lenalidomide on days 1-21, and oral dexamethasone on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with lenalidomide and dexamethasone works in treating patients with relapsed or refractory stage II or stage III multiple myeloma. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab and lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Dexamethasone may stimulate the immune system in different ways and stop cancer cells from growing. Giving bevacizumab together with lenalidomide and dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate (complete response and partial response) in patients with relapsed or refractory stage II or III multiple myeloma treated with bevacizumab, lenalidomide, and dexamethasone.

SECONDARY OBJECTIVES:

I. Determine time to progression in these patients. II. Determine the toxicity and tolerability of this regimen. III. Determine the effect of bevacizumab and lenalidomide on markers of myeloma activity in myeloma cells and stromal cells, including interleukin-6, macrophage inflammatory protein-1α, vascular endothelial growth factor, and STAT3.

IV. Assess local cytokine milieu using tissue microarrays of bone marrow biopsy specimens.

OUTLINE: This is a multicenter, open-label study.

Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, oral lenalidomide on days 1-21, and oral dexamethasone on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and before courses 2 and 4. Blood samples are examined for vascular endothelial growth factor (VEGF) and VEGF receptor (VEGFR) polymorphisms by pyrosequencing and VEGF, VEGFR1, VEGFR2, interleukin-6, and macrophage inflammatory protein 1 by immunoenzyme techniques. Relationships between plasma cell myeloma and stroma and the effect of study treatment on these relationships are examined in tissue sections of bone marrow before and after treatment utilizing microvessel density measurements, VEGF staining, and STAT3 staining (by immunohistochemistry and fluorescent in situ hybridization [FISH]).

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed symptomatic multiple myeloma:

  * Stage II or III disease
  * Relapsed or refractory disease after >= 2 courses of prior chemotherapy
* Measurable levels of monoclonal protein (M protein) > 1.0 g/dL by serum protein electrophoresis OR > 200 mg of monoclonal light chain by 24-hour urine protein electrophoresis
* Measurable bone disease, defined as >= 1 unidimensionally measurable lesion (longest diameter to be recorded) >= 20 mm with conventional techniques OR >= 10 mm with spiral CT scan (for patients with lytic bone disease)
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 70-100%

  * Patients with PS of 3 are eligible if it is due to pain that is likely to improve with treatment
* Life expectancy > 6 months
* No known HIV positivity
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No active infections requiring oral or intravenous antibiotics within the past week
* No proteinuria (i.e., albuminuria) > 1,000 mg/24 hours unless related to the diagnosis of multiple myeloma

  * Patients with light chain (i.e., "Bence-Jones") proteinuria are still eligible if the non-light chain component of protein is < 1,000 mg/24 hours
* No serious nonhealing wound or ulcer
* No blood pressure > 150/90 mm Hg (even with medication)
* No significant traumatic injury within the past 28 days
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No unstable angina or myocardial infarction within the past 6 months
* No stroke within the past 6 months
* No New York Heart Association class III or IV heart failure
* No secondary malignancy within the past 2 years except squamous cell or basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Hemoglobin > 9 g/dL (may be supported by transfusion or growth factors)
* WBC >= 2,000/mm^3
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 75,000/mm^3
* Bilirubin =< 2.5 mg/dL
* At least 4 weeks since prior chemotherapy or radiotherapy and recovered
* More than 7 days since prior minor surgical procedures, fine-needle aspirations, or core biopsies:

More than 24 hours since prior bone marrow biopsy or central veinous access placement

* More than 28 days since prior major surgical procedure or open biopsy
* At least 4 weeks since prior and no concurrent participation in another experimental drug study
* Prior autologous peripheral blood stem cell transplantation allowed
* No prior lenalidomide
* Concurrent full-dose anticoagulants allowed provided all of the following criteria are met:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * No thrombocytopenia requiring transfusion
  * Platelet count > 75,000/mm3
  * INR 2-3 and stable
* No concurrent major surgery
* No concurrent sargramostim (GM-CSF)
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* AST and ALT =< 5 times upper limit of normal
* Creatinine < 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception 4 weeks before, during, and 4 weeks after completion of study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to lenalidomide and/or bevacizumab or other agents used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Callander, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Wisconsin (UW) Hospital and Clinics, the UW 1 South Park Clinic, and the Wisconsin Oncology Network (WON) clinics between November 2006 and March 2011.
Pre-assignment Details: No events between enrollment and group assignment. All subjects enrolled are immediately assigned to Arm 1, "Bevacizumab, Dexamethasone, and Lenalidomide."
Groups:
- Bevacizumab, Dexamethasone, and Lenalidomide: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, oral lenalidomide on days 1-21, and oral dexamethasone on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given IV
  lenalidomide: Given orally
  dexamethasone: Given orally
Period: Overall Study
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Started | 39
Completed | 14
Not Completed | 25
Not completed — Adverse Event | 12
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 5
Not completed — Started Non-Protocol Therapy | 3
Not completed — Stopped treatmen to collect stem cells | 1
Not completed — Transferred to another Institution | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 39
Age, Customized [Number; unit: participants]
  40-49 years | 2
  50-59 years | 4
  60-69 years | 15
  70-79 years | 15
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Anti-tumor Response Rate (Complete Response and Partial Response) to the Combination of Bevacizumab and Lenalidomide
Description: Patient response to the treatment were determined by the definitions for complete response, partial response, marginal response, stable disease, and progressive disease outlined by IMBTR/ABMTR (Blade criteria). Responses were analyzed by descriptive statistics and summarized in tabular format (frequency tables). Furthermore, two-sided 95% confidence intervals for the proportions of subjects with a confirmed anti-tumor response were computed using the method proposed by Chang, which takes into account the multiplicity problem associated with the two-stage testing procedure. The objective response rate was estimated by using Whitehead's bias-adjustment approach.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 39
percentage of participants | 64 [48 to 77]

2. Primary Outcome: Progression Free Survival (Time to Progression)
Description: Patient response to the treatment were determined by the definitions for complete response, partial response, marginal response, stable disease, and progressive disease outlined by IMBTR/ABMTR (Blade criteria). Progression free survival was summarized using point estimates of the median time to progression and associated 95% confidence intervals. The data was presented graphically using Kaplan-Meier plots. Exploratory analysis, including multivariate Cox regression with demographic variables and markers of myeloma activity as covariates was performed.
Time Frame: up to five years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 39
months | 9 [1 to 58]

3. Secondary Outcome: Toxicity and Tolerability of the Bevacizumab and Lenalidomide Combination
Description: Adverse events/toxicities were collected during regular clinical visits. Confidence intervals for the estimate of the true number of patients suffereing from grade 3 or 4 toxicities per common terminology criteria were calculated using the Wilson interval. Ninety-five percent confidence intervals for the proportions of patients with complications (grade 3 or higher toxicities) were constructed.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 39
percentage of participants | 72 [59 to 82]

4. Secondary Outcome: Effect of Bev/Rev on Markers of Myeloma Activity in Myeloma Cells and Stromal Cells at Baseline
Description: A Wilconxon signed-rank test conducted to determine if biomarker levels differed between baseline levels and those after three full cycles of treatment for all patients.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg per liter
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 34
mg per liter
  IL-6 level range | 17.2 (65.1)
  MIP-1 level range | 0.039 (0.025)
  VEGF level range | 0.084 (0.066)
  VEGFR1 level range | 0.12 (0.11)
  VEGFR2 level range | 8.85 (2.08)

5. Secondary Outcome: Local Cytokine Milieu Using Tissue Micro Arrays of Bone Marrow Biopsy Specimens
Time Frame: Up to 5 years
Population: Outcome measure data were not collected.
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 0

6. Secondary Outcome: Effect of Bev/Rev on Markers of Myeloma Activity in Myeloma Cells and Stromal Cells at 3 Months Post-baseline
Description: as for outcome 4
Time Frame: Up to Course 4 Day 1 (3 Months Post-baseline)
Measure: Mean (Standard Deviation); unit: mg per liter
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Number analyzed (Participants) | 34
mg per liter
  IL-6 level range | 5.5 (3.4)
  MIP-1 level range | 0.047 (0.044)
  VEGF level range | 0.054 (0.042)
  VEGFR1 level range | 0.12 (0.088)
  VEGFR2 level range | 8.17 (2.29)

ADVERSE EVENTS:
Arm/Group | Bevacizumab, Dexamethasone, and Lenalidomide
Serious Adverse Events (participants affected / at risk) | 22/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Dexamethasone, and Lenalidomide (N=39)
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Retinal Detachment (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Colonic Perforation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Duodenal Hemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 2
Edema Limbs (General disorders) | 2
Fever (General disorders) | 1
Infections and Infestations, Other (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 2
Mucosal Infection (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Blood Bilirubin Increased (Investigations) | 1
Cardiac Troponin T Increased (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Treatment Related Secondary Malignancy - Chronic Lymphocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysgeusia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic Event (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Dexamethasone, and Lenalidomide (N=39)
Abdominal Pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 4
Alkaline Phosphatase Increased (Investigations) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 21
Anorexia (Metabolism and nutrition disorders) | 14
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8
Blood bilirubin increased (Investigations) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Blurred vision (Eye disorders) | 5
Bruising (Injury, poisoning and procedural complications) | 5
Chills (General disorders) | 4
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Creatinine increased (Investigations) | 6
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 20
Dizziness (Nervous system disorders) | 4
Dry mouth (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Edema limbs (General disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Fatigue (General disorders) | 26
Fever (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 2
Flushing (Vascular disorders) | 3
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Gum infection (Infections and infestations) | 2
Headache (Nervous system disorders) | 11
Hemorrhoids (Gastrointestinal disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 20
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypertension (Vascular disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Hypocalcemia (Metabolism and nutrition disorders) | 17
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 10
Insomnia (Psychiatric disorders) | 9
Lymphocyte count decreased (Investigations) | 15
Mucosal infection (Infections and infestations) | 3
Mucositis oral (Gastrointestinal disorders) | 16
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 10
Neutrophil count decreased (Investigations) | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 15
Personality change (Psychiatric disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Platelet count decreased (Investigations) | 27
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 5
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Tremor (Nervous system disorders) | 5
Upper respiratory infection (Infections and infestations) | 8
Urinary frequency (Renal and urinary disorders) | 2
Urinary Tract Infection (Infections and infestations) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 10
White blood cell decreased (Investigations) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less